CLINICAL TRIAL: NCT05206461
Title: The Trunk Control Which is Fundamental in Hemiparetic and Diparetic Cerebral Palsied Children: Its Relationship With Hand Function and Quality of Life
Brief Title: Relationship Between Trunk Control and Hand Function and Quality of Life
Status: Completed | Type: Observational
Sponsor: KTO Karatay University (Other)
Responsible Party: Sponsor
Other Study IDs: KaratayU1
Record Dates: First submitted 2022-01-11; First posted 2022-01-25 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Cerebral Palsy; Quality of Life; Hand
Keywords: Cerebral Palsy; Trunk Control; Hand Function; Quality of Life
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hemiparetic CP: Trunk control, hand function and quality of life were evaluated with the Trunk Control Measurement Scale, 9-Hole Peg Test and Pediatric Quality of Life Inventory in Hemiparetic CP
  Interventions: Other: Trunk Control Measurement Scale
- Diparetic CP: Trunk control, hand function and quality of life were evaluated with the Trunk Control Measurement Scale, 9-Hole Peg Test and Pediatric Quality of Life Inventory in Diparetic CP
  Interventions: Other: Trunk Control Measurement Scale

INTERVENTIONS:
Other: Trunk Control Measurement Scale — Trunk Control Measurement Scale, easy and simple to use, was used to evaluate trunk control
  Other Names: 9-Hole Peg Test; Pediatric Quality of Life Inventory

SUMMARY:
Increasing quality of life and improving hand functions are very substantial treatment goals for physiotherapy and rehabilitation. Trunk control is important for these parameters in children with hemiparetic and diparetic Cerebral Palsy.

DETAILED DESCRIPTION:
Trunk control, hanf function and quality of life measurements were carried out by a physiotherapist using the Trunk Control Measurement Scale, 9-Hole Peg Test and Pediatric Quality of Life Inventory. Participants were informed about the procedure of the tests. The evaluation period lasted 30-40 minutes for each child.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 5-18,
* Having a diagnosis of hemiparetic or diparetic CP,
* To be at the level of I-II-III according to the Gross Motor Function Classification System,
* Not having had orthopedic surgery on the upper extremity in the last 6 months,
* Not having been injected with Botulinum Toxin-A in the last 6 months,
* Accepting the study and signing the consent form.

Exclusion Criteria:

* Children who could not understand and follow simple verbal commands,
* Did not meet the inclusion criteria,
* Incomplete assessments.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with hemiparetic and diparetic Cerebral Palsy aged 5-18
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-12-13 (Actual)

PRIMARY OUTCOMES:
Trunk Control Measurement Test | Baseline
  Trunk control
9-Hole Peg Test | Baseline
  Hand function
Pediatric Quality of Life Inventory | Baseline
  Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Feride Yarar, Asst Prof,PT, Study Chair — Pamukkale University
Locations (1):
- KTO Karatay University, Konya, Karatay, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No